CLINICAL TRIAL: NCT03797976
Title: The Effects Of Deep Brain Stimulation Of Subthalamıc Nucleus On Pulmonary Function Tests and Functionality In Patıents With Parkinson's Disease: Short Term Results
Brief Title: The Effects Of DBS Of Subthalamıc Nucleus On Functionality In Patıents With Parkinson's Disease: Short-Term Results
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Bircan Yücekaya, Lecturer, Mustafa Kemal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Hatay Mustafa Kemal U 1
Record Dates: First submitted 2018-12-18; First posted 2019-01-09 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Parkinson Disease; Surgery; Respiration; Decreased; Muscle Weakness
MeSH Terms: conditions — Parkinson Disease; Respiratory Insufficiency; Muscle Weakness | interventions — Maximal Respiratory Pressures; Respiratory Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson's Disease Group (Experimental): MIP and MEP Respiratory Function Test Strength Test
  Interventions: Device: MIP and MEP

INTERVENTIONS:
Device: MIP and MEP — Pre-op, Post-op of, 1 month after surgery, 3 months after surgery
  Other Names: Respiratory Function Test; Muscle Test

SUMMARY:
Parkinson's disease is a progressive chronic neurodegenerative disease. In cases where drug treatment is insufficient and drug use is not possible due to drug side effects, highly effective and low-risk surgical treatment options could be used. In Parkinson's Disease; findings such as chest wall rigidity and weakness of the respiratory muscle strength occur. The aim of this study was to determine the effect of preop and postop DBS surgery on respiratory muscle strength, respiratory function and physical performance in patients with Parkinson's disease.

DETAILED DESCRIPTION:
In the study, at least 10 patients with Parkinson's disease who had DBS surgery in Mustafa Kemal University Research and Practice Hospital, Department of Brain and Nerve Surgery will be evaluated. Demographic-physical features, pulmonary functions, respiratory muscle strength, exercise capacity, functionality, and muscle strength will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Lack of any neurological disease other than Parkinson's
* DBS surgery to be performed in the STN region

Exclusion Criteria:

* Patients with advanced cognitive impairment
* Patients with pulmonary, neurological and orthopedic diseases affecting functionalities
* Pregnancy
* Patients in whom the stimulation was canceled due to infection after surgery.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity | Change from Baseline Functional exercise capacity at 3 months(Pre-op,Post-op Off, Post-op 1. month, Post-op 3. Month), an average of 3 months
  6 minute walking test

SECONDARY OUTCOMES:
Pulmonary functions | Change from Pulmonary functions at 3 months(Pre-op,Post-op Off, Post-op 1. month, Post-op 3. Month), an average of 3 months
  Spirometry
Inspiratory and expiratory muscle strength (MIP, MEP) | Change from Inspiratory and expiratory muscle strength (MIP, MEP) at 3 months(Pre-op,Post-op Off, Post-op 1. month, Post-op 3. Month), an average of 3 months
  Mouth pressure device
Muscle strength | Change from Peripheral muscle strength at 3 months(Pre-op,Post-op Off, Post-op 1. month, Post-op 3. Month), an average of 3 months
  Muscle Testing Device (N)
Grip Test (Peripheral muscle strength) | Change from Peripheral muscle strength at 3 months(Pre-op,Post-op Off, Post-op 1. month, Post-op 3. Month), an average of 3 months
  Hand Held Dynamometer (kgf)

CONTACTS AND LOCATIONS:
Overall Officials: Deran Oskay, PhD, Study Director — Gazi University Faculty of Health Science Department of Physical Therapy; Bircan Yucekaya, MSc, Study Chair — Hatay Mustafa Kemal University School of Physical Therapy and Rehabilitation; Atilla Yılmaz, Med. Dr, Principal Investigator — Hatay Mustafa Kemal University Department of Neurosurgery
Locations (1):
- Hatay Mustafa Kemal University, Antakya, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stemper B, Beric A, Welsch G, Haendl T, Sterio D, Hilz MJ. Deep brain stimulation improves orthostatic regulation of patients with Parkinson disease. Neurology. 2006 Nov 28;67(10):1781-5. doi: 10.1212/01.wnl.0000244416.30605.f1. PMID 17130410
- [Background] Trachani E, Constantoyannis C, Sirrou V, Kefalopoulou Z, Markaki E, Chroni E. Effects of subthalamic nucleus deep brain stimulation on sweating function in Parkinson's disease. Clin Neurol Neurosurg. 2010 Apr;112(3):213-7. doi: 10.1016/j.clineuro.2009.11.015. Epub 2009 Dec 22. PMID 20022689
- [Background] Hyam JA, Brittain JS, Paterson DJ, Davies RJ, Aziz TZ, Green AL. Controlling the lungs via the brain: a novel neurosurgical method to improve lung function in humans. Neurosurgery. 2012 Feb;70(2):469-77; discussion 477-8. doi: 10.1227/NEU.0b013e318231d789. PMID 21841525